CLINICAL TRIAL: NCT06158828
Title: A Phase I/II Pilot Study of Memory-like NK Cells to Consolidate TCRαβ T Cell Depleted Haploidentical Transplant in High-risk AML
Brief Title: Pilot Study of Memory-like Natural Killer (ML NK) Cells After TCRαβ T Cell Depleted Haploidentical Transplant in AML
Acronym: ABCD-NK
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Rising Tide Foundation (Other); St. Louis Children's Hospital Foundation (Unknown); Children's' Discovery Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202401147
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: AML, Childhood; Aml; Acute Myeloid Leukemia, Pediatric; Acute Myeloid Leukemia
Keywords: high-risk AML; haploidentical transplant; high-risk acute myeloid leukemia; AML from MDS; memory-like natural killer cells; ML NK cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Antilymphocyte Serum; Busulfan; fludarabine; Thiotepa; Melphalan; Receptors, Antigen, T-Cell, alpha-beta; Interleukin-2; plerixafor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: The study will enroll both transplant recipients and their haploidentical donors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Cohort 1 Recipient: MAC or RIC + Cell graft + ML NK cell infusion (Experimental): * Patients with high-risk genetic features &/or poor response to upfront therapy
  * Myeloablative Conditioning (MAC): rabbit antithymocyte globulin (rATG), Busulfan, Fludarabine, and Thiotepa. All agents are administered intravenously. rATG is administered from days -9 to -7, followed by Busulfan and Fludarabine from days -6 to -3, & Thiotepa on day -2 OR
  * Reduced Intensity Conditioning (RIC): rabbit antithymocyte globulin (rATG), Fludarabine, Melphalan, and Thiotepa. All agents are administered intravenously. rATG is administered from days -9 to -7. Fludarabine is administered from day -8 to day -5, followed by Thiotepa on day -4 and Melphalan on days -3 and -2
  * Patients will undergo infusion of the ex vivo TCRαβ/CD19+ depleted haploidentical HPC graft on day 0. On Day +7, patients will undergo infusion of the memory-like NK (ML NK) cells, followed by IL-2 subcutaneously 4 hours after the infusion. IL-2 will continue every other day through Day +19 for a maximum of 7 doses
- Cohort 2 Recipient: MAC or RIC + Cell graft + ML NK cell infusion (Experimental): * Patients with high-risk AML who meet certain criteria listed in the protocol
  * Myeloablative Conditioning (MAC): rabbit antithymocyte globulin (rATG), Busulfan, Fludarabine, and Thiotepa. All agents are administered intravenously. rATG is administered from days -9 to -7, followed by Busulfan and Fludarabine from days -6 to -3, & Thiotepa on day -2 OR
  * Reduced Intensity Conditioning (RIC): rabbit antithymocyte globulin (rATG), Fludarabine, Melphalan, and Thiotepa. All agents are administered intravenously. rATG is administered from days -9 to -7. Fludarabine is administered from day -8 to day -5, followed by Thiotepa on day -4 and Melphalan on days -3 and -2
  * Patients will undergo infusion of the ex vivo TCRαβ/CD19+ depleted haploidentical HPC graft on day 0. On Day +7, patients will undergo infusion of the memory-like NK (ML NK) cells, followed by IL-2 subcutaneously 4 hours after the infusion. IL-2 will continue every other day through Day +19 for a maximum of 7 doses
- Donor (Other): Donors who meet the eligibility criteria will be mobilized as per institutional standard practice using G-CSF 10 mcg/kg/day for 5 consecutive days. Leukapheresis will be performed after 5 days of G-CSF administration (on Day -1) with a target volume for collection of 20 liters. If additional collection days are necessary to ensure target CD34+ doses, G-CSF administration may be extended per institutional standard and adjusted per physician discretion. Up to 4 days of pheresis are permitted.
  Interventions: Drug: Plerixafor; Biological: Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Rabbit Anti thymocyte globulin — rATG is administered intravenously over 6-18 hours for a total of 2 to 3 doses. The daily dose is based on body weight and lymphocyte count.
  Other Names: rATG
Drug: Busulfan — Busulfan is administered intravenously either Q6H or Q24H, with a recommended target Busulfan AUC of 70-90 mg*h/L.
Drug: Fludarabine — Fludarabine is administered intravenously at a dose of 40 mg/m^2/dose once daily for 4 days.
Drug: Thiotepa — Thiotepa is administered intravenously at a dose of 5 mg/kg/dose Q12H for 2 doses.
Drug: Melphalan — Melphalan is administered intravenously at a dose of 70 mg/m^2/dose once daily for 2 days.
  Other Names: Evolema; Alkeran
Biological: TCR alpha beta / CD19+ depleted haploidentical hematopoietic progenitor cell graft — The HPC product obtained from a haploidentical donor will undergo ex vivo TCR alpha beta and CD19+ depletion, and will be infused fresh on Day 0. There is no maximum limit for CD34+ dose. A maximum dose of 1 x 10^5/kg recipient weight of TCRαβ cells should not be exceeded in the final HPC product.
  Other Names: TCRab/CD19+ depleted haploidentical HPC graft
Biological: memory-like natural killer cells — The ML NK cells (dose: max capped at 20 x 10^6/kg recipient weight, minimum dose allowed is 0.5 x 10^6/kg recipient weight) will be infused on Day +7.
  Other Names: ML NK cells
Biological: IL-2 — IL-2 is administered subcutaneously at a dose of 1 million units/m^2 on Days +7, +9, +11, +13, +15, +17, and +19 (7 doses total).
Drug: Plerixafor — If suboptimal collection of stem cells is predicted, plerixafor may be administered at a dose of 0.24 mg/kg subcutaneous injection once (maximum 40mg/dose). For patients with renal impairment, plerixafor will be administered at a dose of 0.16 mg/kg subcutaneous injection (maximum 27 mg/day).
  Arms: Donor
Biological: Granulocyte Colony-Stimulating Factor — G-CSF will be administered at a dose of 10 mcg/kg/day for 5 days, or 6 days if two days of collection are needed.
  Other Names: G-CSF
  Arms: Donor
Device: CliniMACS — After stem cells are collected by leukapheresis, in order to create the HPC product, the stem cells will be washed to remove platelets and the cell concentration will be adjusted per laboratory and CliniMACS technology recommendations. The cells are then labeled using the CliniMACS TCRαβ Biotin Kit and CD19+ immunomagnetic microbeads. After labeling, the cells are washed to remove unbound microbeads. The partially processed product is loaded on the CliniMACS device where labeled cells are depleted and the negative fraction is eluted off the device. The negative fraction is centrifuged and volume reconstituted to obtain the final product.

SUMMARY:
This trial represents a single institution phase I/II pilot study with the primary objective of establishing the safety and feasibility of generating and infusing ML NK cells after TCRαβ haplo-HCT.

ELIGIBILITY:
Patient Inclusion Criteria - Cohort 1:

1. High risk acute myeloid leukemia (AML) in either:

   1. Complete remission (CR) defined by < 5% marrow blasts by morphology in the context of hematological recovery (ANC ≥ 0.5× 10^9/L, platelet count ≥ 50 × 10^9/L).
   2. Morphological leukemia free state (MLFS) defined by the absence of hematological recovery and < 5% marrow blasts by morphology
2. Patients must further meet one of the below for inclusion into the study:

   1. De novo AML in CR1 with any of the following high-risk features:

      * MRD ≥ 1% after first induction course
      * MRD ≥ 0.1% after second induction course
      * RPN1-MECOM
      * RUNX1-MECOM
      * NPM1-MLF1
      * DEK-NUP214
      * KAT6A-CREBBP (if ≥ 90 days at diagnosis)
      * FUS-ERG
      * KMT2A-AFF1
      * KMT2A-AFDN
      * KMT2A-ABI1
      * KMT2A-MLLT1
      * 11p15 rearrangement (NUP98 - any partner gene)
      * 12p13.2 rearrangement (ETV6 - any partner gene)
      * Deletion 12p to include 12p13.2 (loss of ETV6)
      * Monosomy 5/Del(5q) to include 5q31 (loss of EGR1)
      * Monosomy 7
      * 10p12.3 rearrangement (MLLT10b - any partner gene)
      * FLT3/ITD with allelic ratio > 0.1%, without bZIP CEBPA or NPM1
      * RAM phenotype as evidenced by flow cytometry
      * Other high-risk features not explicitly stated here, after discussion/approval with protocol PI.
   2. De novo AML in ≥ CR2
   3. Therapy-related AML in CR1
   4. AML evolving from myelodysplastic syndrome (MDS)
3. One prior hematopoietic cell transplant is allowed, provided remission criteria as defined above are met.

Patient Inclusion Criteria - Cohort 2:

1. High risk acute myeloid leukemia (AML) defined by either of the following:

   1. Treatment refractory disease: AML that is not in complete remission despite prior standard or salvage therapies.
   2. Multiply relapsed disease: AML that has relapsed after 2 or more hematopoietic cell transplantations.
2. BM disease burden: Less than 25% bone marrow blasts by morphology must be present (M2 marrow), irrespective of peripheral hematological recovery.

Patient Inclusion Criteria - Both Cohorts:

1. Less than or equal to 40 years of age.
2. Lansky (<16 years) or Karnofsky (≥16 years) performance status of >60%.
3. Adequate organ function as defined below:

   1. Total bilirubin ≤ 3 x IULN for age
   2. AST(SGOT)/ALT(SGPT) ≤ 5 x IULN for age
   3. GFR ≥ 60 mL/min/1.73m2 as estimated by (1) updated Schwartz formula for ages 1-17 years or Cockcroft-Gault formula for ages ≥ 18 years, (2) 24-hour creatinine clearance, or (3) renal scintigraphy. If GFR is abnormal for age based on updated Schwartz or Cockcroft-Gault formula, accurate measurement should be obtained by either 24-hour creatinine clearance or renal scintigraphy.
   4. Renal function may also be estimated by serum creatinine based on age/gender. A serum creatinine < 2 x IULN for age/gender is required for inclusion on this protocol.
4. Adequate cardiac function, defined by left ventricular ejection fraction (LVEF) at rest ≥50% or shortening fraction (SF) ≥27% (via echocardiogram or MUGA).
5. Adequate pulmonary function, defined by:

   1. FEV1, FVC, and DLCO ≥50% of predicted.
   2. O2 saturation ≥ 92% on room air by pulse oximetry and no supplemental O2 at rest for children < 8 years of age or those unable to perform pulmonary function testing (PFT). For children unable to perform PFT, a high-resolution CT chest should be obtained.
6. The effects of these treatments on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 24 months following transplant. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
7. Ability to understand and willingness to sign an IRB approved written informed consent document, or patient has a guardian who has the ability to understand and willingness to sign an IRB approved written informed consent document.
8. Available familial haploidentical donor. The HCT donor must be available and willing to undergo 2 leukapheresis procedures: (I) one mobilized collection for the HPC graft and (II) one non-mobilized leukapheresis collection for the manufacturing of ML NK cells.
9. Donor and recipient must be identical at a minimum of one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA- DQB1. A minimum of 5/10 match is required and will be considered sufficient evidence that the donor and recipient share one HLA haplotype.

Patient Exclusion Criteria - Both Cohorts

1. Active GvHD. If patient had prior GvHD, patient must be off immunosuppression for at least 3 months prior to starting study treatment.
2. Active non-hematologic malignancy. History of other malignancy is acceptable as long as therapy has been completed and there is no current evidence of disease.
3. Currently receiving any other investigational agents at the time of transplant.
4. Active CNS or extramedullary disease. History of CNS or extramedullary disease currently in remission is acceptable.
5. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study.
6. Inability to discontinue medications that are likely to interfere with ML NK cell activity, i.e., glucocorticoids and other immunosuppressants.
7. Presence of significant anti-donor HLA antibodies per institutional standards. Anti-donor HLA - Antibody Testing is defined as a positive crossmatch test of any titer (by complement dependent cytotoxicity or flow cytometric testing) or the mean fluorescence intensity (MFI) of any anti-donor HLA antibody by solid phase immunoassay > 3000.
8. Presence of a second major disorder deemed a contraindication for HCT.
9. Patients with Fanconi Anemia or Down Syndrome.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (bacterial, viral with clinical instability, or fungal), symptomatic congestive heart failure, or unstable cardiac arrhythmia.
11. Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of the start of conditioning.

Donor Eligibility Criteria - Both Cohorts

1. Donor must be at least 18 years of age.
2. Donor must be HLA haploidentical (≥ 5/10 and ≤ 9/10 allele match at the -A, -B, -C, DRB1 and DQ loci) by high resolution typing and related to the patient.
3. Donor must meet the selection criteria as defined by the Foundation for the Accreditation of Hematopoietic Cell Therapy (FACT).
4. Donor must be available and willing to undergo one mobilized and one non-mobilized leukapheresis procedure.
5. Donor may not be pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days prior to initiation of recipient's conditioning regimen, within 7 days of donor stem cell mobilization regimen and prior to second non-mobilized leukapheresis..
6. Donor must be able to understand and willing to sign an IRB-approved written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety of patients being administered donor-derived ML NK cells following TCR alpha beta depleted haploidentical cell transplant | From transplant through Day +100
  Safety will be determined by events occurring following transplant. Non-relapse mortality, engraftment failure, and development of severe GvHD will be considered events.
Feasibility of manufacturing and administering donor-derived ML NK cells following TCR alpha beta depleted haploidentical cell transplant | Through time of ML NK cell infusion (around Day +7)
  Feasibility is defined by product manufacture failure, i.e., the inability to infuse ML NK cells due to product contamination or insufficient cell dose (<0.5x10^6 / kg recipient weight).

SECONDARY OUTCOMES:
Relapse Free Survival (RFS) | From transplant through Month 12
  Defined as the time between the date of transplant and date of last follow up, relapse, or death due to any cause.
Overall Survival (OS) | From transplant through Month 12
  Defined as death from any cause following transplant.
Development of acute graft versus host disease (aGvHD) | From transplant through Day +100
  Incidence of grade II, III, or IV acute GvHD as graded according to the NIH consensus criteria. Severe aGvHD (Grades III-IV) is considered an event.
Development of chronic graft versus host disease (cGvHD) | From transplant through Day +180
  Incidence of chronic GvHD as graded according to the NIH consensus criteria. Severe cGvHD is considered an event.
Development of chronic graft versus host disease (cGvHD) | From transplant through Day +365
  Incidence and severity of chronic GvHD as graded according to the NIH consensus criteria. Severe cGvHD is considered an event.
Development of infections | From transplant through Day +180
  Significant infections include, but are not limited to, bacterial or fungal sepsis, viral reactivation with or without clinical disease, other viral infections, and community acquired infections.
Analysis of immune reconstitution | From transplant through Month 24
  Immune reconstitution is defined as regain of function of donor-derived immunogenic cells and is measured by recovery of individual cellular compartments.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Pfeiffer, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu